CLINICAL TRIAL: NCT01397435
Title: Quantification of Bone Marrow Involvement in Gaucher Disease With Proton MR Spectroscopy, Correlation With Bone Marrow Burden Score, Genotype and Disease Severity Score for Pediatric Patients
Brief Title: MR Spectroscopy and Disease Severity Score for Gaucher in Pediatric Population
Acronym: MRS in Gaucher
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-008013
Record Dates: First submitted 2011-06-13; First posted 2011-07-19 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Gaucher
Keywords: Lysosomal diseases; Magnetic resonance Spectroscopy; MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gaucher: We will enroll 15 children who have a confirmed diagnosis of Gaucher disease.
- Healthy volunteers: We will enroll 15 age and gender matched controls.

SUMMARY:
The bone status in Gaucher disease is very difficult to monitor precisely in children. This is a major problem because lack of optimal treatment, especially enzyme replacement, may cause irreversible severe bone damage that will impact an affected person's life. Currently, there are qualitative (subjective) methods, such as Magnetic resonance Imaging (MRI), to gauge the response to treatment. A quantitative (objective) measurement of Gaucher cell presence and activity in bone marrow could help with more precise and accurate monitoring of bone marrow disease in patients both treated and not (yet) being treated with enzyme replacement. The investigators will evaluate the efficacy of Magnetic Resonance Spectroscopy (MRS) as a quantitative assessment of bone marrow involvement in Children with Gaucher, and examine how this result correlates with semiquantitative MRI scales and overall disease severity.

DETAILED DESCRIPTION:
To quantify the amount of fat in the bone marrow of affected subjects and healthy controls the investigators will use Single voxel short, echo time(TE) proton spectroscopy. This MR Spectroscopy (MRS) will be conducted in the vertebral body of L5 and in the neck of the femur.

To assess the qualitative scores and compare it to the quantitative MR Spectroscopy (MRS) results the investigators will use a series of Fluid sensitive and Fat sensitive conventional MR sequences that will allows us to determine indirectly the degree of glucocerebrosidase infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Gaucher disease / age and gender match control
* Children aged 5-20 yrs
* Parental consent
* Child assent if appropriate

Exclusion Criteria:

* Presence of medical illness or exposure to drugs that alter the appearance of bone marrow on MRI
* Contraindication for MRI
* Likelihood for claustrophobia
* Non cooperative patient
* Pregnancy

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will enroll patients with a Diagnosis of Gaucher disease. Subjects will be between 5 and 20 years of age. We will recruit an equal number of age and gender matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference in the fat fraction (quantified by MRS) between subjects with Gaucher disease and controls. | within 5 minutes
  We will measure the fat fraction only once, at the time of recruitment. We will compare the fat fraction of an affected subject to that of an age matched control. We will determine if significant difference exist.

SECONDARY OUTCOMES:
Difference in the semiquantitative MRI scores between affected subjects and controls | within 5 minutes
  We will compare the ordinal data obtained from applying two semiquantitative severity scores: Bone marrow burden (BMB) and Spanish MRI (S-MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Jaramillo, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia; Paige Kaplan, MBBCh, Study Chair — Children's Hospital of Philadelphia; Maria A Bedoya, MD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Kaplan P, Andersson HC, Kacena KA, Yee JD. The clinical and demographic characteristics of nonneuronopathic Gaucher disease in 887 children at diagnosis. Arch Pediatr Adolesc Med. 2006 Jun;160(6):603-8. doi: 10.1001/archpedi.160.6.603. PMID 16754822
- [Background] Maas M, van Kuijk C, Stoker J, Hollak CE, Akkerman EM, Aerts JF, den Heeten GJ. Quantification of bone involvement in Gaucher disease: MR imaging bone marrow burden score as an alternative to Dixon quantitative chemical shift MR imaging--initial experience. Radiology. 2003 Nov;229(2):554-61. doi: 10.1148/radiol.2292020296. Epub 2003 Oct 2. PMID 14526090
- [Background] Charrow J, Andersson HC, Kaplan P, Kolodny EH, Mistry P, Pastores G, Rosenbloom BE, Scott CR, Wappner RS, Weinreb NJ, Zimran A. The Gaucher registry: demographics and disease characteristics of 1698 patients with Gaucher disease. Arch Intern Med. 2000 Oct 9;160(18):2835-43. doi: 10.1001/archinte.160.18.2835. PMID 11025794
- [Background] Roca M, Mota J, Alfonso P, Pocovi M, Giraldo P. S-MRI score: A simple method for assessing bone marrow involvement in Gaucher disease. Eur J Radiol. 2007 Apr;62(1):132-7. doi: 10.1016/j.ejrad.2006.11.024. Epub 2006 Dec 11. PMID 17161930
- [Background] Weinreb NJ, Cappellini MD, Cox TM, Giannini EH, Grabowski GA, Hwu WL, Mankin H, Martins AM, Sawyer C, vom Dahl S, Yeh MS, Zimran A. A validated disease severity scoring system for adults with type 1 Gaucher disease. Genet Med. 2010 Jan;12(1):44-51. doi: 10.1097/GIM.0b013e3181c39194. PMID 20027115
- [Background] Maas M, Hangartner T, Mariani G, McHugh K, Moore S, Grabowski GA, Kaplan P, Vellodi A, Yee J, Steinbach L. Recommendations for the assessment and monitoring of skeletal manifestations in children with Gaucher disease. Skeletal Radiol. 2008 Mar;37(3):185-8. doi: 10.1007/s00256-007-0425-0. No abstract available. PMID 18094966
- [Background] Baldellou A, Andria G, Campbell PE, Charrow J, Cohen IJ, Grabowski GA, Harris CM, Kaplan P, McHugh K, Mengel E, Vellodi A. Paediatric non-neuronopathic Gaucher disease: recommendations for treatment and monitoring. Eur J Pediatr. 2004 Feb;163(2):67-75. doi: 10.1007/s00431-003-1363-z. Epub 2003 Dec 16. PMID 14677062